CLINICAL TRIAL: NCT06924177
Title: Utilizing Dietician-guided Intervention to Combat Neurogenic Obesity in People With Spinal Cord Injury
Brief Title: UTSW NORC Pilot Spinal Cord Injury Dietary Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Yi-Ting Tzen, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU20250145
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Obesity-related Medical Conditions; Spinal Cord Injury, Chronic
Keywords: spinal cord injuries; obesity; insulin resistance
MeSH Terms: conditions — Obesity; Spinal Cord Injuries; Bronchiolitis Obliterans Syndrome; Insulin Resistance | interventions — Telemedicine; Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experiment (Experimental): 9 weeks of Telehealth with dietician using DPP modules diet portion. The nine modules are:
  1. Eat well to prevent T2DM
  2. Track your food
  3. Shop and cook to prevent T2DM
  4. Eat well away from home
  5. Stay motivated to prevent T2DM
  6. More about carbs
  7. Have health food you enjoy
  8. Get back on track
  9. Prevent T2DM for life
  Interventions: Other: Telehealth with dietician

INTERVENTIONS:
Other: Telehealth with dietician — 9 weeks of telehealth visit with dietician using the DPP diet modules

SUMMARY:
The goal of this observational study is to learn about the effects of a 9-week dietician-guided program modified from the National Diabetic Prevention Program (modified DPP-diet) in people with spinal cord injury on body composition and insulin sensitivity.

The main question it aims to answer is:

Does 9 week modified DPP-diet reduce body fat percentage and insulin resistance?

Participants will:

Have 9 weeks of Telehealth visit with dietician certified in providing DPP. Visit the laboratory before, immediately and 9 weeks after completion of the modified DPP-diet.

Share with the researcher on the perceived benefit and obstacles in implementing the modified DPP-diet as part of their daily activities.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years old
* have had SCI for more than one year
* not independently ambulatory
* primarily uses a wheelchair for mobility
* community-dwelling
* without comorbidities listed in the exclusion criteria

Exclusion Criteria:

* uncontrolled type 2 diabetes mellitus
* pregnancy
* active systemic disease, e.g., heart disease, real failure/insufficiency, multiple myeloma, lupus with nephropathy, sickle cell disease, symptomatic myasthenia gravis, poorly controlled hypo- or hyperthyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
body fat composition | from enrollment to 9 weeks after completion of the modified DPP-diet program
  Whole body fat percentage from dual-energy X-ray absorptiometry scan. The unit will be %, with higher value indicating larger amount of body fat within an individual.
Homeostatic Model Assessment 2 for Insulin Resistance (HOMA2-IR) | from enrollment to 9 weeks after completion of the modified DPP-diet program
  An insulin resistance index calculated from fasting glucose (mmol/l) and insulin (μU/ml) level from blood draw. The HOMA2-IR will be calculated using the formula: HOMA2-IR = (Fasting Insulin (μU/ml) * Fasting Glucose (mmol/L)) / 22.5.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
age, gender, body mass index, whole body fat percentage, HOMA2-IR value
Supporting Information: Study Protocol
Time Frame: 12/31/2026-12/31/2030
Access Criteria: Any researchers interested in the data could reach out to the PI directly with a proposal to request the data. Data will be shared de-identified.